CLINICAL TRIAL: NCT02364271
Title: Improving Early Risk Stratification in Patients Presenting to Emergency Departments With Undifferentiated Chest Pain
Brief Title: Early Risk Stratification in ED Chest Pain Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Timothy H Rainer, Director & Professor, Chinese University of Hong Kong
Other Study IDs: 10110121
Record Dates: First submitted 2015-02-03; First posted 2015-02-18 (Estimated); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Acute Coronary Syndrome
Keywords: High-sensitive troponin; TIMI score; Major adverse cardiac event; HEART score
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Fibrinolytic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Not low risk for MACE in 30 days: Patients with not low risk of major adverse cardiac events within 30 days Patients with TIMI>0 or mHEART>2
  Routine blood test for hs-cTnT and Thrombolysis in myocardial infarction (TIMI) score were performed on study patients
  Protocol amendment:
  In October 2014, mHEART score of the study patients was determined retrospectively
  Interventions: Other: Thrombolysis in myocardial infarction score; Biological: routine blood test for hs-cTnT; Other: HEART score
- Low risk for MACE in 30 days: Patients with low risk of major adverse cardiac events within 30 days
  Patients with TIMI=0 and mHEART<=2
  Routine blood test for hs-cTnT and Thrombolysis in myocardial infarction (TIMI) score were performed on study patients
  Protocol amendment:
  In October 2014, mHEART score of the study patients was determined retrospectively
  Interventions: Other: Thrombolysis in myocardial infarction score; Biological: routine blood test for hs-cTnT; Other: HEART score

INTERVENTIONS:
Other: Thrombolysis in myocardial infarction score — An English- and Cantonese-speaking research nurse obtained the TIMI scores which consists of seven variables from each eligible patient.
  Other Names: TIMI score
Biological: routine blood test for hs-cTnT — Patient had routine venipuncture blood taking for hs-cTnT measurement in the central laboratory of the hospital. Normal level of hs-cTnT is below 14ng/L.
  Other Names: hs-cTnT
Other: HEART score — The modified HEART score of each patient was determined retrospectively by a research assistant.

SUMMARY:
In the management of adult chest pain patients presenting to an Emergency Department (ED) with suspected acute coronary syndrome (ACS), we aimed to evaluate the diagnostic accuracy of the combined use of a modified Thrombolysis in Myocardial Infarction (TIMI) score and a modified HEART score with high-sensitive cardiac troponin T (hs-cTnT) to rule out major adverse cardiac events (MACE) in 30-days.

DETAILED DESCRIPTION:
Chest pain is one of the most common complaints in patients presenting to emergency departments (ED) globally, representing 2.5% of all ED presentations in Hong Kong. Acute coronary syndrome (ACS) cannot be immediately excluded in the majority of patients presenting with chest pain, and is confirmed in about 15-25% cases. The current evaluation of patients in most EDs is a lengthy process that involves serial ECGs and troponin tests taken 3-6 hours apart. However, challenges over ED crowding and the need for acceptable risk stratification have prompted the search for safe, cheap, but effective accelerated chest pain pathways.

An ever increasing evidence base is emerging from emergency departments in different geographical settings, using different combinations of clinical assessment tools, more rapid biochemical tests and variable outcomes. While making an accurate diagnosis is clearly important, from the patients' perspective it is more important to minimize the risk of adverse events. Therefore, the identification of tools which allow risk stratification to permit very low risks of MACE is more clinically relevant to ED specialists than the precise diagnostic label applied to the patient.

In the Asia-Pacific region a 2-hour diagnostic protocol involving serial point-of-care biomarkers, such as troponin I, creatine kinase MB, and myoglobin, combined with electrocardiograph (ECG) changes and a Thrombolysis in Myocardial Infarction (TIMI) score has been shown to safely exclude 30-day MACE in low risk patients with chest pain. Highly sensitive troponin T (hs-cTnT) and troponin I (hs-cTnI) perform well in the early diagnosis of acute myocardial infarction (AMI), non-ST elevation myocardial infarction (NSTEMI) and in the prediction of two year mortality. Undetectable levels of hs-cTnT alone at initial blood testing appears to rule-out 60-day NSTEMI with a negative predictive value of 94% and a sensitivity of 90%. A TIMI score incorporating hs-cTnT was no better at predicting 30-day MACE than front-door TIMI alone without measurement of biomarkers, but the value of a TIMI score of zero in ruling-out low risk patients was not demonstrated.

Despite evidence favouring early rule out pathways, there is still a need for further validation and refinement of such tools using different diagnostic pathways, in other clinical settings, and with other clinical tools such as HEART.

In this study we aimed firstly to evaluate the effectiveness of a combined use of an early modified TIMI score with hs-cTnT and a modified HEART score to rule out MACE in 30 days. Applying this protocol in clinical practice has the potential to reduce ED waiting times, ED crowding and hospital admission rates for chest pain patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Chest pain within 24 hours of ED presentation
* Suspected with ACS

Exclusion Criteria:

* No cardiac chest pain based on clinical assessment
* Hemodynamic or clinical instability (SBP<90 mmHg, clinically significant atrial/ventricular arrhythmias)
* Initial ECG suggestive of ACS, Acute Myocardial Infarction or other abnormality requiring admission to hospital
* Previous coronary artery bypass grafting or coronary stent implantation
* Women with known or suspected pregnancy
* Unable or unwilling to provide informed consent
* Unable to be contacted after discharge
* Contraindication to β-blockade if prescription of β-blockade is required due to a resting heart rate over 80 beats per minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had chest or epigastric pain within 24 hours of emergency department presentation and suspected with acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H Rainer, MD FCEM, Principal Investigator — Accident & Emergency Medicine Academic Unit
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Background] Pope JH, Aufderheide TP, Ruthazer R, Woolard RH, Feldman JA, Beshansky JR, Griffith JL, Selker HP. Missed diagnoses of acute cardiac ischemia in the emergency department. N Engl J Med. 2000 Apr 20;342(16):1163-70. doi: 10.1056/NEJM200004203421603. PMID 10770981
- [Background] Chou KL, Chow NW, Chi I. Preventing economic hardship among Chinese elderly in Hong Kong. J Aging Soc Policy. 2004;16(4):79-97. doi: 10.1300/J031v16n04_05. PMID 15724574
- [Background] Bernstein SL, Aronsky D, Duseja R, Epstein S, Handel D, Hwang U, McCarthy M, John McConnell K, Pines JM, Rathlev N, Schafermeyer R, Zwemer F, Schull M, Asplin BR; Society for Academic Emergency Medicine, Emergency Department Crowding Task Force. The effect of emergency department crowding on clinically oriented outcomes. Acad Emerg Med. 2009 Jan;16(1):1-10. doi: 10.1111/j.1553-2712.2008.00295.x. Epub 2008 Nov 8. PMID 19007346
- [Background] Viswanathan K, Kilcullen N, Morrell C, Thistlethwaite SJ, Sivananthan MU, Hassan TB, Barth JH, Hall AS. Heart-type fatty acid-binding protein predicts long-term mortality and re-infarction in consecutive patients with suspected acute coronary syndrome who are troponin-negative. J Am Coll Cardiol. 2010 Jun 8;55(23):2590-8. doi: 10.1016/j.jacc.2009.12.062. PMID 20513600
- [Background] Kilcullen N, Viswanathan K, Das R, Morrell C, Farrin A, Barth JH, Hall AS; EMMACE-2 Investigators. Heart-type fatty acid-binding protein predicts long-term mortality after acute coronary syndrome and identifies high-risk patients across the range of troponin values. J Am Coll Cardiol. 2007 Nov 20;50(21):2061-7. doi: 10.1016/j.jacc.2007.08.021. Epub 2007 Nov 5. PMID 18021874
- [Background] Nabi F, Chang SM, Pratt CM, Paranilam J, Peterson LE, Frias ME, Mahmarian JJ. Coronary artery calcium scoring in the emergency department: identifying which patients with chest pain can be safely discharged home. Ann Emerg Med. 2010 Sep;56(3):220-9. doi: 10.1016/j.annemergmed.2010.01.017. Epub 2010 Feb 6. PMID 20138399
- [Background] Blaha MJ, Budoff MJ, DeFilippis AP, Blankstein R, Rivera JJ, Agatston A, O'Leary DH, Lima J, Blumenthal RS, Nasir K. Associations between C-reactive protein, coronary artery calcium, and cardiovascular events: implications for the JUPITER population from MESA, a population-based cohort study. Lancet. 2011 Aug 20;378(9792):684-92. doi: 10.1016/S0140-6736(11)60784-8. PMID 21856482
- [Background] Antman EM, Cohen M, Bernink PJ, McCabe CH, Horacek T, Papuchis G, Mautner B, Corbalan R, Radley D, Braunwald E. The TIMI risk score for unstable angina/non-ST elevation MI: A method for prognostication and therapeutic decision making. JAMA. 2000 Aug 16;284(7):835-42. doi: 10.1001/jama.284.7.835. PMID 10938172
- [Background] Conway Morris A, Caesar D, Gray S, Gray A. TIMI risk score accurately risk stratifies patients with undifferentiated chest pain presenting to an emergency department. Heart. 2006 Sep;92(9):1333-4. doi: 10.1136/hrt.2005.080226. No abstract available. PMID 16908715
- [Background] Mettler FA Jr, Huda W, Yoshizumi TT, Mahesh M. Effective doses in radiology and diagnostic nuclear medicine: a catalog. Radiology. 2008 Jul;248(1):254-63. doi: 10.1148/radiol.2481071451. PMID 18566177
- [Background] Rumberger JA, Brundage BH, Rader DJ, Kondos G. Electron beam computed tomographic coronary calcium scanning: a review and guidelines for use in asymptomatic persons. Mayo Clin Proc. 1999 Mar;74(3):243-52. doi: 10.4065/74.3.243. PMID 10089993
- [Background] Chan CP, Sum KW, Cheung KY, Glatz JF, Sanderson JE, Hempel A, Lehmann M, Renneberg I, Renneberg R. Development of a quantitative lateral-flow assay for rapid detection of fatty acid-binding protein. J Immunol Methods. 2003 Aug;279(1-2):91-100. doi: 10.1016/s0022-1759(03)00243-6. PMID 12969550
- [Background] Miller CD, Lindsell CJ, Anantharaman V, Lim SH, Greenway J, Pollack CV, Tiffany BR, Hollander JE, Gibler WB, Hoekstra JW; EMCREG-International i*trACS Investigators. Performance of a population-based cardiac risk stratification tool in Asian patients with chest pain. Acad Emerg Med. 2005 May;12(5):423-30. doi: 10.1197/j.aem.2004.11.016. PMID 15863398
- [Background] Kip KE, Hollabaugh K, Marroquin OC, Williams DO. The problem with composite end points in cardiovascular studies: the story of major adverse cardiac events and percutaneous coronary intervention. J Am Coll Cardiol. 2008 Feb 19;51(7):701-7. doi: 10.1016/j.jacc.2007.10.034. PMID 18279733
- [Background] Liao J, Chan CP, Cheung YC, Lu JH, Luo Y, Cautherley GW, Glatz JF, Renneberg R. Human heart-type fatty acid-binding protein for on-site diagnosis of early acute myocardial infarction. Int J Cardiol. 2009 Apr 17;133(3):420-3. doi: 10.1016/j.ijcard.2008.01.049. Epub 2008 Jun 20. PMID 18571749
- [Background] Chan CP, Sanderson JE, Glatz JF, Cheng WS, Hempel A, Renneberg R. A superior early myocardial infarction marker. Human heart-type fatty acid-binding protein. Z Kardiol. 2004 May;93(5):388-97. doi: 10.1007/s00392-004-0080-6. PMID 15160274
- [Background] Six AJ, Cullen L, Backus BE, Greenslade J, Parsonage W, Aldous S, Doevendans PA, Than M. The HEART score for the assessment of patients with chest pain in the emergency department: a multinational validation study. Crit Pathw Cardiol. 2013 Sep;12(3):121-6. doi: 10.1097/HPC.0b013e31828b327e. PMID 23892941

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Low Risk Group: Routine blood test for hs-cTnT, Thrombolysis in myocardial infarction score (TIMI) and mHEART score were performed on study patients. TIMI>0 and mHEART>2
- Low Risk Group: Routine blood test for hs-cTnT, Thrombolysis in myocardial infarction score (TIMI) and mHEART score were performed on study patients. TIMI=0 or mHEART<=2
Period: Overall Study
Arm/Group | Not Low Risk Group | Low Risk Group
Started | 479 | 123
Completed | 479 | 123
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Risk Group: Routine blood test for hs-cTnT, Thrombolysis in myocardial infarction score (TIMI) and mHEART score were performed on study patients. TIMI>0 and mHEART>2
- Total: Total of all reporting groups
Arm/Group | High Risk Group | Low Risk Group | Total
Number analyzed (Participants) | 479 | 123 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 165 | 116 | 281
  >=65 years | 314 | 7 | 321
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.5 [57.5 to 78] | 66 [56 to 78] | 66 [56 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 67 | 308
  Male | 238 | 56 | 294
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 479 | 123 | 602
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 42 | 560 | 602

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Major Adverse Cardiac Event
Description: The primary outcome is the number of patients with MACE within 30 days after initial ED presentation. MACE is defined as relating to safety outcome, or effecacy outcome.
Time Frame: 30 days
Population: This is not an interventional trial. This prospective observational study to assess the efficiency of combining TIMI and HEART score in early exclusion of major adverse cardiac events in emergency department patients with chest pain
Measure: Count of Participants; unit: Participants
Groups:
- Not Low Risk Groups: Patients with modified TIMI>0 and modified HEART>2 were considered as high risk for 30-day MACE.
  Modified TIMI and HEART scores included hs-cTnT tests as opposed to conventional cTnT in the original tests. The presence of any ST-deviation of >0.05mV in the initial ECG was considered a positive result. A negative hs-cTnT result was defined as a concentration of ≤14ng/L.
- Low Risk Group: Patients with modified TIMI=0 or modified HEART<=2 were considered as low risk for 30-day MACE.
  Modified TIMI and HEART scores included hs-cTnT tests as opposed to conventional cTnT in the original tests. The presence of any ST-deviation of >0.05mV in the initial ECG was considered a positive result. A negative hs-cTnT result was defined as a concentration of ≤14ng/L.
Arm/Group | Not Low Risk Groups | Low Risk Group
Number analyzed (Participants) | 479 | 123
Participants
  MACE within 30 days | 42 | 0
  No MACE within 30 days | 437 | 123

2. Secondary Outcome: Number of Safety Major Adverse Cardiac Event
Description: Outcome is the number of patients with safety MACE within 30 days after initial ED presentation. Safety MACE is defined as relating to safety outcome,which consists of all-cause mortality (included cardiac death),cardiac arrest,readmission with myocardial infarction and cardiogenic shock
Time Frame: 30 Days
Population: Patients with major adverse cardiac events occurred within 30-days
Measure: Count of Participants; unit: Participants
Groups:
- Not Low Risk Group: Patients with modified TIMI>0 and modified HEART>2 were considered as high risk for 30-day MACE.
  Modified TIMI and HEART scores included hs-cTnT tests as opposed to conventional cTnT in the original tests. The presence of any ST-deviation of >0.05mV in the initial ECG was considered a positive result. A negative hs-cTnT result was defined as a concentration of ≤14ng/L.
Arm/Group | Not Low Risk Group | Low Risk Group
Number analyzed (Participants) | 42 | 0
Participants | 31 | 0

3. Secondary Outcome: Number of Effecacy MACE
Description: Outcome is the number of patients with effecacy MACE within 30 days after initial ED presentation. Effecacy MACE consists of revascularization (e.g.coronary artery bypass grafting),ventricular arrhythmia needing intervention and high-degree atrioventricular block needing intervention.
Time Frame: 30 days
Population: Patient had MACE within 3 months of initial presentation for chest pain in ED
Measure: Count of Participants; unit: Participants
Arm/Group | Not Low Risk Group | Low Risk Group
Number analyzed (Participants) | 42 | 0
Participants | 26 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Major adverse cardiac events encompass both safety and effecacy elements. Safety outcomes consist of all-cause mortality (including cardiac death), cardiac arrest, myocardial infarction and cardiogenic shock. Effecacy outcomes consist of revascularization (e.g. coronary artery bypass grafting or percutaneous coronary intervention), ventricular arrhythmia needing intervention and high-degree atrioventricular block needing intervention
Groups:
- Not Low Risk Group: Patients with modified TIMI>0 and modified HEART>2 were considered as high risk for 30-day MACE.
- Low Risk Group: Patients with modified TIMI=0 or modified HEART<=2 were considered as low risk for 30-day MACE.
Arm/Group | Not Low Risk Group | Low Risk Group
All-Cause Mortality (participants affected / at risk) | 5/479 | 0/123
Serious Adverse Events (participants affected / at risk) | 26/479 | 0/123
Other Adverse Events (participants affected / at risk) | 9/479 | 0/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Low Risk Group (N=479) | Low Risk Group (N=123)
Safety MACE (STEMI) (Cardiac disorders) | 10 (10) | 0 (0) — Patients had STEMI and survived. 7 had percutaneous coronary intervention or coronary artery bypass grafting
Safety MACE (NSTEMI) (Cardiac disorders) | 16 (16) | 0 (0) — Patients had NSTEMI and survived. 10 had percutaneous coronary intervention or coronary artery bypass grafting
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Low Risk Group (N=479) | Low Risk Group (N=123)
Effectiveness MACE (PCI) (Surgical and medical procedures) | 7 (7) | 0 (0) — Percutaneous coronary intervention without prior serious adverse cardiac event.
Effectiveness MACE (CABG) (Surgical and medical procedures) | 2 (2) | 0 (0) — Coronary artery bypass grafting without prior serious adverse cardiac event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No